CLINICAL TRIAL: NCT06412276
Title: Out-of-home Consumer Food Purchase Behaviour in the Presence and Absence of Value Pricing and Price Promotions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool John Moores University (Other); University of Bristol (Other); Economic and Social Research Council, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Price-based incentive study
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-05

CONDITIONS: Food Selection; Healthy Eating; Eating Behavior
MeSH Terms: conditions — Food Preferences; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: participants will be randomly assigned to one of five conditions.
Who Masked: Participant
Masking Description: Participants will not know the treatment group to which they have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control (Experimental): Food menu typical for the out-of-home outlet with
  * Product price promotions (25% off orders over £10)
  * Bulk buy reductions (bundle options for reduced prices)
  * Volume value pricing (increase in size for a disproportionately small increase in price)
  Interventions: Behavioral: Control
- Product price reductions removed (Experimental): Food menu without product price promotions
  Interventions: Behavioral: Product price promotions removed
- Bulk buy price reductions removed (Experimental): Food menu without price decrease for bulk-buy items (i.e. bundles available but not at a decreased price)
  Interventions: Behavioral: Bulk buy reductions removed
- Volume value pricing removed (Experimental): For products on the food menu with size increases, increases in price will be made proportionate (as opposed to value)
  Interventions: Behavioral: Volume value pricing removed
- No price-based incentive (Experimental): Food menus will be provided with no price-based incentives
  Interventions: Behavioral: No price-based incentives

INTERVENTIONS:
Behavioral: Control — Food menu will be provided as is typical for the out of home outlet
  Arms: Control
Behavioral: Product price promotions removed — Food menus with no price reductions to products
  Arms: Product price reductions removed
Behavioral: Bulk buy reductions removed — Food menus with bundles provided but not at reduced prices
  Arms: Bulk buy price reductions removed
Behavioral: Volume value pricing removed — Food menus with proportionate pricing for multi-size products
  Arms: Volume value pricing removed
Behavioral: No price-based incentives — Food menus with no price-based incentives offered
  Arms: No price-based incentive

SUMMARY:
It is important to understand the role that price-based incentives in the out-of-home food sector play in food purchasing, and whether they lead to positive savings for the consumer (as they would likely anticipate when making purchases), or whether these incentives lead to increased spending and increased purchasing of unhealthy products. Additionally, it is important to consider whether the impacts of price-based incentives differ according to a range of demographic characteristics. For example, some evidence suggests that effects of removing a price-based incentive are greater in individuals with a higher BMI. Evidence also suggests there may also be differences in impact according to socioeconomic position (SEP) as individuals in lower SEP groups reportedly use price-based incentives more frequently. If lower SEP individuals are more affected by price-based incentives (i.e. they prompt ordering in excess and greater spend), then the banning of such strategies could help to reduce health inequalities, by nudging lower SEP consumers toward healthier dietary choices in the OOH food sector.

To date, it is unclear what effect policies which remove specific types of price-based incentives would be likely to have on consumer behaviour. In particular, individual product price reductions (e.g. £ off this product), bulk buy price reductions (e.g., Save £ when bought together) and volume value pricing (e.g., the price increase from a small to large portion size not being directly proportional to volume increase).

Therefore our primary objectives are:

• To observe the effect of removing price-based incentives (individual product price reductions, bulk buy price reductions, volume value pricing) in the OOH food sector on:

* Energy purchased per household
* Money spent per household

Secondary Objectives:

• To explore whether any effects of removing price-based incentives differ based on participant characteristics (BMI, SEP, food choice motives)

DETAILED DESCRIPTION:
See attached study protocol for detailed information

ELIGIBILITY:
Inclusion Criteria:

* Currently reside in the United Kingdom
* Over the age of 18 years
* Fluent English speaker Frequently use food delivery apps or websites (at least once a month, on average)
* Frequently eat takeaway pizza (i.e. once every 2-3 months)
* Can complete the study on a laptop or desktop

Exclusion Criteria:

* Partaking in a fast or other restrictive eating for religious reasons at time of participation
* Dietary restrictions/intolerances including:

  * Gluten-free
  * Dairy-free
  * Sugar-free

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2051 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Energy (kcal) ordered | immediately after food choice
  The total energy content of the hypothetical food order
Monetary value of order | immediately after food choice
  The total monetary value of the hypothetical food order
Likelihood of using a bulk-buy promotion | immediately after food choice
  The likelihood of participants selecting a bulk-buy option or 'bundle'
Likelihood of selecting a larger or smaller size | immediately after food choice
  The likelihood of participants selecting a larger or smaller size for food items with multi-size options

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study data (anonymised) will be shared on the Open Science Framework (OSF)
Supporting Information: Study Protocol, SAP
Time Frame: On publication, indefinitely
Access Criteria: Open website
URL: https://osf.io/fxc8q/?view_only=9ee32fbe61ef4a26bb4fb7662dacc7d1